CLINICAL TRIAL: NCT06657495
Title: Thử Nghiệm Lâm Sàng Giai Đoạn 2, Ngẫu Nhiên, Mù Đôi, Có Đối Chứng Giả Dược Để Đánh Giá Tính an Toàn Và Hiệu Quả Của Viên Hoàn Cứng TD0015 Trên Bệnh Nhân Thoái Hóa Khớp Gối
Brief Title: To Evaluate the Safety and Efficacy of TD0015 Pilulae in Patients with Knee Osteoarthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sao Thai Duong Joint Stock Company (Industry)
Collaborators: Big Leap Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TD0015
Record Dates: First submitted 2024-09-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Three arms: basic dose, 1.5 basic dose and placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo pilulae weighing 5g/pack, after a meal, 1pack/time x 2 times/day
  Interventions: Drug: TD0015 Placebo
- Investigational product 1 (Experimental): estimated dose:TD0015 pilulae weighing 5g/pack , after a meal, 1pack/time x 2 times/day
  Interventions: Drug: TD0015
- Investigational product 2 (Experimental): 1.5 times of estimated dose: TD0015 pilulae weighing 7.5g/pack , after a meal, 1pack/time x 2 times/day
  Interventions: Drug: TD0015

INTERVENTIONS:
Drug: TD0015 — TD0015 is black, dark brown inside pilulae and has special smell of herbal, slightly sour then bitter taste.
  Arms: Investigational product 1; Investigational product 2
Drug: TD0015 Placebo — Placebo was packed in pack 5g
  Arms: Placebo

SUMMARY:
Preclinical trials in animal models have suggested that the estimated dose of TD0015 in clinical presents no safety concerns.The investigational product is TD0015 pilulae, which is based on the traditional prescription named "Độc hoạt tang ký sinh thang" (Thien Kim Phuong).

The traditional prescription has the effect of circulating blood in the tendons and bones to bring out evil spirits, blood tonic, kidney tonic to prevent recurrence of diseases and against joint degeneration, joint deformation, muscle atrophy, stiffness to recover normal joint function.

DETAILED DESCRIPTION:
The study objective is to evaluate the safety and efficacy of TD0015 pilulae to determine the optimal dose for investigational product. Phase II analyzes is performed on 90 patients and based on the results of phase II to adjust sample size and study design (if applicable) for phase III.

The trial lasts for ~ 30 months with 6 subject visits (from T0 to T5) and is conducted in National Hospital of Traditional Medicine (Hanoi, Vietnam).

Screening procedure occurs at T0 visit, followed by T1 (15+/-3 days), T2 (30+/-3 days), T3 (45+/-3 days), T4 (60+/-3 days) and T5 (90+/-3 days). The telephone contact visits are performed every 2 weeks by Investigators There are 2 levels of dosages: estimated dose - 5g (arm 1) and 1.5 times (arm 2) of estimated dose - 7.5g. There is also another arm using placebo, thus the trial have 3 arms in total.

As for 3 arms, patients is allowed to use oral NSAIDs (meloxicam 7,5mg x 1-2 tablets/day) when pain is severe.

Treatment time is 60 days. IP is used after a meal, 1 pack/time x 2 times/day.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients ≥ 18 years old must meet ALL or the following criteria clusters 1,2,6 or 1,3,5,6 or 1,4,5,6 to be enrolled:

1. Knee pain
2. Bone spurs forming along the edges of the joint, narrowing of joint space in X-ray film (grade I-III) according to Kellgren and Lawrence
3. Knee joint effusion
4. Morning stiffness that lasts less than 30 minutes when moving
5. Knee crepitus when moving
6. Patient voluntarily agree and and sign in the ICF

According to traditional medicine: The disease type is Wind-Cold-Damp Bi with Kidney and Liver Deficiency. Symptoms are knee joint is pain, cold and heavy. Pain is usually fixed, little movement, mild during the day, severe at night, increased in cold and wet weather. Warm compresses to relieve pain, knee joint may be swollen, limited movement, may have morning stiffness, joint deformity associated with muscle atrophy, back pain, not warm limbs.The tongue is pale, the tongue is white and greasy, and deep-thready-weak pulse.

Exclusion Criteria:

1. Hypersensitivity to any subtances of TD0015 pilulae.
2. Pregnant or lactating
3. Currently having surgical indications.
4. Other conditions asseted by the investigator that are not eligible to be enrolled.
5. Knee Osteoarthritis grade IV according to classification of Kellgren and Lawrence (specify that large osteophytes, marked narrowing of joint space, severe sclerosis and definite deformity of bone ends)
6. Self-administration of other anti-inflammatory medicine (except for NSAIDs) during study period as for 3 arms
7. Patient is treated by NSAIDs within 3 days or has corticosteroid Intra-articular injection within 3 months prior to enrolment
8. Joint and/or systemic infections
9. Cardiovascular diseases (arrhythmia, hypertension) without treatment
10. Cross - hypertensitivity to aspirin or other NSAIDs
11. History of recent or progressive peptic ulcer/gastrointestinal perforation
12. Severe liver failure
13. Severe renal failure without dialysis
14. Gastrointestinal hemorrhage, recent brain hemorrhage or disorders causing systemic hemorrhage
15. Uncontrolled heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on the Western Ontario and McMaster Universities Osteoarthrities Index) WOMAC to evaluate the level of symptoms | Day 15th, day 30th, day 45th, day 60th and day 30th after end of study
  WOMAC was scored by investigator in visits (T1, T2, T3, T4, T5) and compared with T0
Change from baseline in Pain Scores on the Visual Analog Scale | day 15th, day 30th, day 45th, day 60th and day 30th after end of study
  VAS scale: 0 = no pain | 0-->2: mild | 2-->4: moderate | 4--> 6: severe | 6->8: extreme | 8-->10: untolerable
  Evaluate outcome of treatment according to VAS scale:
  * Very Good: 0
  * Good: 1 - 4
  * Average: 5 - 7
  * Weak: >8
Change in symptoms severity was reported by patient on the Lequesne Index | day 15th, day 30th, day 45th, day 60th and day 30th after end of study
  Lequesne Index at prior and after treatment (day 15th, day 30th, day 45th, day 60th and day 30th after end of study).
Percentage of patients taking rescue medication | 90 days
  3 Arms were allowed to use oral NSAIDs (meloxicam 7,5 mg x 1-2 tablets/day) when pain was severe. All NSAIDs in the study need to be documented in detail
The average dose of rescue medication was used | 90 days
Frequency of AE, SAE | 90 days
  Reference CTCAE 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital of Traditional Medicine, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ha NTT, Nghia DT, Nga HTV, Lua TT, Hong NTB, Hanh NT, Ngoc NK, Vuong NL. Traditional Vietnamese herbal medicine TD0015 in Knee Osteoarthritis: A Phase-II randomized controlled trial. Integr Med Res. 2025 Jun;14(2):101143. doi: 10.1016/j.imr.2025.101143. Epub 2025 Mar 31. PMID 40290409